CLINICAL TRIAL: NCT06901687
Title: Home-Based tDCS for Depression in Multiple Sclerosis: A Randomized Sham-Controlled Trial
Brief Title: Home-Based Transcranial Direct Current Stimulation (tDCS) for Depression in Multiple Sclerosis (MS)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 25-00165
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Multiple Sclerosis; Depression
Keywords: Multiple Sclerosis; Depression; Neuromodulation; Home-Based; transcranial direct current stimulation
MeSH Terms: conditions — Multiple Sclerosis; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active tDCS (Experimental): Participants will complete 30 x 30 minute daily (M-F) sessions of active tDCS which will be paired with a mindfulness meditation audio track.
  Interventions: Device: Active tDCS
- Sham tDCS (Sham Comparator): Participants will complete 30 x 30 minute daily (M-F) sessions of sham tDCS which will be paired with a mindfulness meditation audio track.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — tDCS is a noninvasive brain stimulation technique that delivers a low-intensity electrical current (2.0 mA) through sponge electrodes placed on the scalp. For Active tDCS, the device is programmed to ramp up to 2.0 mA (for 30 seconds), provide constant current throughout session (29 minutes), and then ramp down (for 30 seconds) at the end.
  Arms: Active tDCS
Device: Sham tDCS — tDCS is a noninvasive brain stimulation technique that delivers a low-intensity electrical current (2.0 mA) through sponge electrodes placed on the scalp. For Sham tDCS (or placebo) the device is programmed to ramp up to 2.0 mA (for 30 seconds) followed by a ramp down (30 seconds), with no current delivery for 28 minutes, and then ramp up (for 30-s) and down (for 30-s) at the end.
  Arms: Sham tDCS

SUMMARY:
This project is a double-blind, sham-controlled, parallel-arm, randomized controlled trial. We will recruit n=170 people living with MS, who are experiencing an episode of depression in the context of a major depressive episode (MDE). Using our remotely supervised (RS) tDCS protocol, enrolled participants will complete 30 days of 30-minute tDCS (2.0, DLPFC left anodal) while listening to mindfulness meditation. Over the course of the study, participants will complete assessments of depression and MS symptoms. Participants will be randomized 1:1 active:sham tDCS.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years (inclusive)
* Diagnosis: Confirmed diagnosis of multiple sclerosis (MS), including relapsing-remitting or secondary progressive subtypes
* Stable Medications: Stable use of antidepressant and disease-modifying therapies (DMTs) for at least 30 days prior to enrollment
* Stable Disease Activity: Defined as no clinical relapse, no new radiological disease activity, and no recent steroid treatment for at least 30 days prior to enrollment
* Provider Contact: Confirmed access to a local provider that has primary responsibility for the subjects' clinical care, and who is available for contact in case of increased subject risk due to depressive symptoms
* Technical Ability: Ability to use mobile devices and participate in remote, video-supervised sessions

Exclusion Criteria:

* Neurological or Medical Disorders: History of primary neurological disorder other than MS (e.g., stroke, Parkinson's disease, traumatic brain injury (TBI), intracranial mass, epilepsy, mild cognitive impairment (MCI), dementia), major psychiatric disorders (e.g., bipolar disorder, psychotic disorders), or serious medical conditions (e.g., myocardial infarction, thyroid disease, diabetes with complications, atrial fibrillation)
* Substance Use: Nicotine use (e.g., smoking or vaping) within the past 6 months
* Pregnancy and Breastfeeding: Currently pregnant, planning pregnancy during the study period, or breastfeeding. If able to become pregnant, participants will be required to use medically accepted birth control methods, including hormonal methods (e.g., pills, patches, implants), barrier methods (e.g., condoms or diaphragm with spermicide), intrauterine device (IUD), or abstinence. Participants will be advised not to become pregnant during the study.
* Seizure History: History of seizures or seizure disorder within the past 5 years
* Implanted Devices or Metal Objects: Presence of metal in the head/neck area (excluding dental fillings) or implanted medical devices (e.g., neurostimulators, pacemakers, defibrillators)
* Skin Conditions: Active skin disorders or skin sensitivity near electrode application sites

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Hamilton Depression Rating Scale (HDRS-17) | Baseline, Week 8 (End of Intervention)
  HDRS-17 is a 17-item assessement of depression symptoms. Each item is rated on a Likert scale; the total score is the sum of responses and ranges from 0-52, with higher scores indicating greater levels of depression. A score of 0-7 is generally accepted to be within the normal range (or in clinical remission), while a score of 20 or higher indicates at least moderate severity.
Change in Hamilton Depression Rating Scale (HDRS-17) | Baseline, Month 3
  HDRS-17 is a 17-item assessement of depression symptoms. Each item is rated on a Likert scale; the total score is the sum of responses and ranges from 0-52, with higher scores indicating greater levels of depression. A score of 0-7 is generally accepted to be within the normal range (or in clinical remission), while a score of 20 or higher indicates at least moderate severity.

SECONDARY OUTCOMES:
Change in SymptoMScreen Score | Baseline, Week 8 (End of Intervention)
  12-item measure of overall MS symptom burden. Each item is rated on a scale from 0 (not affected at all) to 6 (total limitation). The total score is the sum of responses and ranges from 0 to 72; higher scores indicate greater overall MS symptom burden.
Change in SymptoMScreen Score | Baseline, Month 3
  12-item measure of overall MS symptom burden. Each item is rated on a scale from 0 (not affected at all) to 6 (total limitation). The total score is the sum of responses and ranges from 0 to 72; higher scores indicate greater overall MS symptom burden.
Change in Cognitive Processing Speed (SDMT) | Baseline, Week 8 (End of Intervention)
  The Symbol Digit Modalities Test (SDMT) scores the total number of correct symbol-digit substitutions within 90 seconds, with a higher score indicating better cognitive processing speed. The maximum possible score is 110, the minimum possible score is 0.
Change in Cognitive Processing Speed (SDMT) | Baseline, Month 3
  The Symbol Digit Modalities Test (SDMT) scores the total number of correct symbol-digit substitutions within 90 seconds, with a higher score indicating better cognitive processing speed. The maximum possible score is 110, the minimum possible score is 0.
Change in Quality of Life in Neurological Disorders (Neuro-QOL) Scale v1.0 - Communication Score | Baseline, Week 8 (End of Intervention)
  Neuro-QOL Scale - Communication Subscale comprises 5 items assessing respondents' difficulty in performing everyday tasks requiring communication. Each item is rated on a scale from 1 (cannot perform) to 5 (no difficulty). The total score is the sum of responses and ranges from 5-25; higher scores indicate greater communication abilities function.
Change in Quality of Life in Neurological Disorders (Neuro-QOL) Scale v1.0 - Communication Score | Baseline, Month 3
  Neuro-QOL Scale - Communication Subscale comprises 5 items assessing respondents' difficulty in performing everyday tasks requiring communication. Each item is rated on a scale from 1 (cannot perform) to 5 (no difficulty). The total score is the sum of responses and ranges from 5-25; higher scores indicate greater communication abilities function.
Proportion of Participant who Achieve Clinical Response per HDRS-17 at End of Intervention | Week 8 (End of Intervention)
  Clinical response is defined as a ≥ 50% reduction in HDRS-17 score from baseline to end of intervention.
Proportion of Participant who Achieve Clinical Response per HDRS-17 at Month 3 Follow-Up | Month 3
  Clinical response is defined as a ≥ 50% reduction in HDRS-17 score from baseline to end of intervention.
Proportion of Participant who Achieve Remission per HDRS-17 at End of Intervention | Week 8 (End of Intervention)
  Clinical response is defined as a HDRS-17 score ≤ 7 at the end of intervention.
Proportion of Participant who Achieve Remission per HDRS-17 at Month 3 Follow-Up | Month 3
  Clinical response is defined as a HDRS-17 score ≤ 7 at the end of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Charvet, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
At this time, there are no plans to share Individual Participant Data (IPD) due to considerations related to participant confidentiality, data security, and the study's intended scope. However, summary-level findings will be disseminated through publications and presentations.